CLINICAL TRIAL: NCT01151852
Title: A Prospective, Double Blind, Randomized, Placebo-Controlled Phase III Trial of Imatinib Re-Challenge in Patients With Gastrointestinal Stromal Tumor Who Had Benefit From Prior Imatinib But Progression From Both Imatinib and Sunitinib
Brief Title: Rechallenge of Imatinib in GIST Having no Effective Treatment: RIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Study Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMC1001
Record Dates: First submitted 2010-06-23; First posted 2010-06-29 (Estimated); Results first posted 2015-07-28 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Imatinib; Re-challenge
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imatinib (Experimental): Patients will be randomly assigned to receive imatinib at a dose of 400mg/day, taken once daily with food, in the form of 100-mg tablets. The study medication will be administered until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Imatinib
- Placebo (Placebo Comparator): Patients will be randomly assigned to receive placebo at a dose of 400mg/day, taken once daily with food, in the form of 100-mg tablets. The study medication will be administered until disease progression or withdrawal of consent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imatinib — Patients will be randomly assigned to receive imatinib at a dose of 400mg/day, taken once daily with food, in the form of 100-mg tablets. The study medication will be administered until disease progression, unacceptable toxicity, or withdrawal of consent.
  Other Names: Glivec
  Arms: Imatinib
Drug: Placebo — Patients will be randomly assigned to receive placebo at a dose of 400mg/day, taken once daily with food, in the form of 100-mg tablets. The study medication will be administered until disease progression or withdrawal of consent.
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the clinical outcomes following resumption of dosing (re-challenge) with Imatinib plus best supportive care versus placebo plus best supportive care in patients with advanced/incurable Gastrointestinal Stromal Tumors following failure of prior imatinib and sunitinib therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients with metastatic or unresectable malignant gastrointestinal stromal tumour which has been histologically confirmed by the detection of CD117 on immunohistochemical staining or genetically confirmed by the detection of mutation in KIT or PDGFRα genes on direct sequencing of tumor DNA.
* Prior benefit from 1st line imatinib defined as complete response, partial response, or stable disease at 6 months after the start of 1st line imatinib
* Patients whose disease has progressed despite at least both prior imatinib therapy (400mg/day) and then subsequently also failure of prior sunitinib therapy.
* ECOG(Eastern Cooperative Oncology Group) performance status 0 ~ 3
* Adequate bone marrow function as defined by platelets ≥ 75 x 109/L and neutrophils ≥ 1.5 x 109/L
* Adequate renal function, with serum creatinine < 1.5 x upper limit of normal
* Adequate hepatic function with serum total bilirubin < 1.5 x upper limit of normal, alanine aminotransferase or aspartate aminotransferase < 2.5 x upper limit of normal in the absence of liver metastases, or < 5 x upper limit of normal in the presence of liver metastases.
* Expected life expectancy of greater than 12 weeks in the absence of any intervention
* No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other cancer except where treated with curative intent > 5 years previously without evidence of relapse
* Written, informed consent to the study

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol or a history of non- compliance
* Last dose of radiotherapy received within 4 weeks before the start of study treatment, excluding palliative radiotherapy
* Obstruction of gastrointestinal tract
* Active gastrointestinal bleeding
* Myocardial infarction within 6 months prior to the study medication, and other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol
* Female patients who are pregnant or breast-feeding. Female patients must have had a negative pregnancy test within one week before starting imatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Background] Corless CL, Fletcher JA, Heinrich MC. Biology of gastrointestinal stromal tumors. J Clin Oncol. 2004 Sep 15;22(18):3813-25. doi: 10.1200/JCO.2004.05.140. PMID 15365079
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Demetri GD, von Mehren M, Blanke CD, Van den Abbeele AD, Eisenberg B, Roberts PJ, Heinrich MC, Tuveson DA, Singer S, Janicek M, Fletcher JA, Silverman SG, Silberman SL, Capdeville R, Kiese B, Peng B, Dimitrijevic S, Druker BJ, Corless C, Fletcher CD, Joensuu H. Efficacy and safety of imatinib mesylate in advanced gastrointestinal stromal tumors. N Engl J Med. 2002 Aug 15;347(7):472-80. doi: 10.1056/NEJMoa020461. PMID 12181401
- [Background] De Giorgi U, Verweij J. Imatinib and gastrointestinal stromal tumors: Where do we go from here? Mol Cancer Ther. 2005 Mar;4(3):495-501. doi: 10.1158/1535-7163.MCT-04-0302. PMID 15767559
- [Background] Verweij J, Casali PG, Zalcberg J, LeCesne A, Reichardt P, Blay JY, Issels R, van Oosterom A, Hogendoorn PC, Van Glabbeke M, Bertulli R, Judson I. Progression-free survival in gastrointestinal stromal tumours with high-dose imatinib: randomised trial. Lancet. 2004 Sep 25-Oct 1;364(9440):1127-34. doi: 10.1016/S0140-6736(04)17098-0. PMID 15451219
- [Background] Debiec-Rychter M, Sciot R, Le Cesne A, Schlemmer M, Hohenberger P, van Oosterom AT, Blay JY, Leyvraz S, Stul M, Casali PG, Zalcberg J, Verweij J, Van Glabbeke M, Hagemeijer A, Judson I; EORTC Soft Tissue and Bone Sarcoma Group; Italian Sarcoma Group; Australasian GastroIntestinal Trials Group. KIT mutations and dose selection for imatinib in patients with advanced gastrointestinal stromal tumours. Eur J Cancer. 2006 May;42(8):1093-103. doi: 10.1016/j.ejca.2006.01.030. Epub 2006 Apr 18. PMID 16624552
- [Background] Demetri GD, van Oosterom AT, Garrett CR, Blackstein ME, Shah MH, Verweij J, McArthur G, Judson IR, Heinrich MC, Morgan JA, Desai J, Fletcher CD, George S, Bello CL, Huang X, Baum CM, Casali PG. Efficacy and safety of sunitinib in patients with advanced gastrointestinal stromal tumour after failure of imatinib: a randomised controlled trial. Lancet. 2006 Oct 14;368(9544):1329-38. doi: 10.1016/S0140-6736(06)69446-4. PMID 17046465
- [Derived] Yoo C, Ryu MH, Nam BH, Ryoo BY, Demetri GD, Kang YK. Impact of imatinib rechallenge on health-related quality of life in patients with TKI-refractory gastrointestinal stromal tumours: Sub-analysis of the placebo-controlled, randomised phase III trial (RIGHT). Eur J Cancer. 2016 Jan;52:201-8. doi: 10.1016/j.ejca.2015.10.071. Epub 2015 Dec 14. PMID 26699729
- [Derived] Kang YK, Ryu MH, Yoo C, Ryoo BY, Kim HJ, Lee JJ, Nam BH, Ramaiya N, Jagannathan J, Demetri GD. Resumption of imatinib to control metastatic or unresectable gastrointestinal stromal tumours after failure of imatinib and sunitinib (RIGHT): a randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1175-82. doi: 10.1016/S1470-2045(13)70453-4. Epub 2013 Oct 18. PMID 24140183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 20, 2010, and Jan 17, 81 patients were enrolled in Asan Medical Center, Seoul, Korea.
Pre-assignment Details: Randomization was done in a double-blind manner and stratified by performance status (0-1 vs 2-3) and by the number of previous lines of tyrosine-kinase inhibitor therapy (2 or less vs more than 2).
Period: Overall Study
Arm/Group | Imatinib | Placebo
Started | 41 | 40
Completed | 41 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Our analysis was based on intention-to treat population. So, all enrolled patients were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib | Placebo | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 25 | 54
  >=65 years | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.4) | 59.6 (10.6) | 58.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 29 | 26 | 55
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: To compare the progression free survival (PFS) assessed by the blinded independent central review following resumption of dosing (re-challenge) with Imatinib plus best supportive care versus placebo plus best supportive care in patients with unresectable or metastatic GIST following failure of at least prior imatinib and sunitinib therapies
Time Frame: up tp12 weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 41 | 40
Months | 1.8 [1.7 to 3.6] | 0.9 [0.9 to 1.7]

2. Secondary Outcome: Disease Control Rate
Description: Inclusion of complete response, partial response or stable disease
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Progressive disease (PD), >20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), Insufficient change to qualify for PR or PD.
Time Frame: up to 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 41 | 40
percentage of participants | 32 | 5

3. Secondary Outcome: Progression Free Survival
Description: To compare PFS assessed by investigators
Time Frame: up to 12 weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 41 | 40
Months | 1.8 [1.7 to 2.7] | 1.7 [0.9 to 1.8]

4. Secondary Outcome: Response Rate
Description: Tumour responses were initially determined by the local investigators in accordance with RECIST 1.0.Treatment decisions were based on local onsite radiological review. All imaging data were subsequently collected, anonymised, and reviewed centrally in a double-blind manner by two external academic radiology reviewers.
  Response assessment was determined in a masked central review by use of RECIST1.1.
Time Frame: Up to 12weeks
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 41 | 40
percentage of participants | 0 | 0

5. Secondary Outcome: Overall Survival(OS) and Time to Progression(TTP)
Description: To compare the overall survival (OS) and time to progression (TTP) in both arms of the study
Time Frame: Up to 3years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 41 | 40
Months
  Overall survival | 8.2 [5.5 to 12.8] | 7.5 [4.4 to 12.4]
  Time to progression | 1.8 [1.7 to 3.6] | 0.9 [0.9 to 1.7]

6. Secondary Outcome: Safety and Tolerability of Imatinib
Description: percentage of patients who experienced toxicity from study treatment to evaluate the safety and tolerability of imatinib re-challenge in this patient population
Time Frame: Up to 3years
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib | Placebo
Number analyzed (Participants) | 41 | 40
percentage of participants | 100 | 98

ADVERSE EVENTS:
Arm/Group | Imatinib | Placebo
Serious Adverse Events (participants affected / at risk) | 1/41 | 2/40
Other Adverse Events (participants affected / at risk) | 41/41 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=41) | Placebo (N=40)
Edema (Musculoskeletal and connective tissue disorders) | 1 | 0 — Grade 3 edema
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Grade 3 diarrhea
Vomiting (Gastrointestinal disorders) | 0 | 1 — Grade 3 vomiting
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (N=41) | Placebo (N=40)
Neutropenia (Blood and lymphatic system disorders) | 12 | 5
Anemia (Blood and lymphatic system disorders) | 27 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 3
Edema (Musculoskeletal and connective tissue disorders) | 18 | 5
Fatigue (General disorders) | 15 | 5
Anorexia (Gastrointestinal disorders) | 14 | 8
Nausea (Gastrointestinal disorders) | 13 | 1
Vomiting (Gastrointestinal disorders) | 13 | 2
Constipation (Gastrointestinal disorders) | 6 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 4
Hyperbilirubinemia (Hepatobiliary disorders) | 10 | 6
Azotemia (Renal and urinary disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No